CLINICAL TRIAL: NCT05386719
Title: A Cardiometabolic Screening Program for Breast Cancer Survivors
Brief Title: Cardiometabolic Screening Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Private Philanthropic Funds (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: J21125; IRB00285627 (Other: Johns Hopkins Medicine)
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Early-stage Breast Cancer
Keywords: Survivor
MeSH Terms: conditions — Breast Neoplasms | interventions — Mass Screening; BaseLine dental cement; Health Planning Guidelines

STUDY DESIGN:
Intervention Model Description: The screening program will refer patients to established institutional programs and resources (Cardiovascular Disease prevention program, Healthful Weight Eating Activity Program and Endocrinology).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early stage breast cancer survivors (Other): Patients with history of early stage breast cancer and at least 3 months from completion of local and systemic therapy at Johns Hopkins
  Interventions: Other: Prescreening; Other: Screening and Enrollment; Behavioral: Baseline; Behavioral: Interpret BMI; Other: Interpret HbA1c; Other: Interpret lipid panel and assess other risk factors; Behavioral: Assess 10 year risk of cardiovascular event; Behavioral: Recommendations; Behavioral: Follow-Up

INTERVENTIONS:
Other: Prescreening — Eligible patients (history of early stage breast cancer and at least 3 months from completion of local and systemic therapy at Johns Hopkins, reads and speaks English) complete survey for demographics, smoking status & questions about cardiovascular disease.
Other: Screening and Enrollment — Consent
Behavioral: Baseline — Behavioral Battery and Patient Reported Outcome Quality of Life questionnaires (EORTC QLQ-C30 and QLQ-BR23) Labs (Hba1c + lipid panel if not done within 12 months or if abnormal within 1 year) Abstract vitals from chart review
  Other Names: Patient- reported outcomes questionnaires, labs, vitals results
Behavioral: Interpret BMI — Refer to Healthful Eating, Activity and Weight Program (HEAWP) if BMI ≥25 and not already on lifestyle intervention
Other: Interpret HbA1c — HbA1c results categorized as follows:
  HbA1c <5.7%; HbA1c 5.7-6.4%; HbA1c 6.5%+; or Known diabetic on medication
Other: Interpret lipid panel and assess other risk factors — Based on above categories:
  HbA1c <5.7%: Any of these cardiovascular disease risk factors: current/former tobacco use, total cholesterol >200, family history of Coronary Artery Disease/Heart Attack in first degree family <55 year old male or <65 year old female, systolic blood pressure >130 HbA1c 5.7-6.4%: Refer to Primary Care Provider and consider Healthful Eating, Activity and Weight Program (HEAWP) HbA1c 6.5%+: Refer to Endocrinology if HbA1c ≥8% Known diabetic on medication: Refer to Endocrinology if HbA1c ≥7%
Behavioral: Assess 10 year risk of cardiovascular event — If risk factors are present - refer to Cardiovascular Disease Prevention Program
Behavioral: Recommendations — Provide individual patient handout based on all above interventions
Behavioral: Follow-Up — 6 and 12 month labs (if prior abnormal) and Patient Reported Outcome questionnaires

SUMMARY:
This research study is being done to implement a screening program for prediabetes, diabetes, dyslipidemia and/or hyperlipidemia, and higher risk of cardiovascular disease in breast cancer survivors. This program will also help to direct individuals with risk factors to community and institutional resources for management.

DETAILED DESCRIPTION:
The investigators propose a prospective cardiometabolic screening program for breast cancer survivors. A formalized screening program may ensure that all patients are receiving these routine screening tests. This program could not only serve to detect prediabetes, diabetes, dyslipidemia and/or hyperlipidemia, but also direct individuals with other risk factors to community and institutional resources for management.

HYPOTHESIS

* Prediabetes, diabetes, dyslipidemia and overweight/obesity are prevalent in women with early stage breast cancer.
* Participants that continue to participate in the study will have lower HbA1c, lower LDL, percent weight loss, and change in patient-reported outcomes (quality of life, function and symptoms) at 6 and 12 months compared to baseline.
* Risk factors for cardiovascular disease (such as tobacco use, family history, hypertension) are common in breast cancer patients.
* The screening program will refer patients to established institutional programs and resources (Cardiovascular Disease prevention program, Healthful Weight Eating Activity Program and Endocrinology).
* The prevalence of prediabetes, diabetes and dyslipidemia in women with breast cancer will be significantly higher than healthy controls from a national database, matched for age and other comorbidities.

OBJECTIVES

Primary Objectives

1. To estimate the prevalence of prediabetes, diabetes, dyslipidemia and overweight/obesity in women with early stage breast cancer
2. To estimate the proportion of participants with lower HbA1c, lower LDL, percent weight loss, and change in patient-reported outcomes (quality of life, function and symptoms) at 6 and 12 months compared to baseline.

Secondary Objectives

1. To estimate the prevalence of other risk factors for cardiovascular disease (tobacco use, family history, hypertension) in breast cancer patients
2. To report the number of referrals of individuals with diabetes or prediabetes or risk factors for cardiovascular disease (CVD) to established institutional programs and resources.
3. To compare the prevalence of prediabetes, diabetes and dyslipidemia in women with breast cancer with healthy controls from a national database, matched for age and other comorbidities.

Exploratory

1. To assess change in HbA1c from baseline 6 and 12 months, and use of antidiabetes pharmacotherapy for patients referred to Endocrinology for diabetes management
2. To assess change in total cholesterol and LDL from baseline to 6 and 12 months, and use of statins, aspirin or antihypertensives for patients referred to CVD prevention program
3. To assess percent weight loss, and use of pharmacotherapy in patients referred to institutional weight loss program

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of early stage breast cancer
* Completed local and/or systemic therapy at least 3 months ago
* Receiving medical oncology care at through the breast cancer clinics at Johns Hopkins Medical Institute, including the Sidney Kimmel Comprehensive Cancer Center in Baltimore MD and Green Spring Station in Lutherville-Timonium MD, and Sibley Memorial Hospital in Washington D.C.
* Read and speak English

Exclusion Criteria:

* Metastatic breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of prediabetes | 3 years
  The proportion of women with early stage breast cancer who have prediabetes: The number is determined through medical history, laboratory results, and baseline survey. Prevalence of prediabetes, will be estimated with an exact 95% confidence interval.
Prevalence of diabetes | 3 years
  The proportion of women with early stage breast cancer who have diabetes: The number is determined through medical history, laboratory results, and baseline survey. Prevalence of diabetes, will be estimated with an exact 95% confidence interval.
Prevalence of hyperlipidemia | 3 years
  The proportion of women with early stage breast cancer with hyperlipidemia as determined by medical history and laboratory results. Prevalence of hyperlipidemia will be estimated with an exact 95% confidence interval.
Change in HbA1c | Baseline, 6 months, 12 months
  The percent change in HbA1c laboratory results, at 6 and 12 months compared to baseline.
Change in LDL cholesterol | Baseline, 6 months, 12 months
  The percent change in LDL cholesterol (mg/dL) laboratory results at 6 and 12 months compared to baseline.
Prevalence of obesity/ overweight | Baseline, 6 months, 12 months
  The proportion of women with early stage breast cancer with BMI >/= 25kg/mg squared. Body Mass Index (BMI) as recorded in participant electronic medical record will be evaluated to determine the percent change in Body Mass Index from baseline at 6 and 12 months.
Quality of Life Questionnaire The European Organisation for Research and Treatment Cancer C30 | Baseline, 6 months, 12 months
  Participants will complete the Quality of Life Questionnaire C30 The Quality of Life Questionnaire-C30, which includes 30 items. The 30 items assess physical, role, emotional, cognitive and social functioning, global health status or Quality Of Life scales, fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties. The Quality of Life Questionnaire-C30 is scored on the basis of classical test theory (CTT), and uses the total item score as the scale score. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient). The percent change in Patient Reported Outcome scores from baseline is accessed at 6 months and 12 months.
Breast-specific symptoms assessed by the of The European Organisation for Research and Treatment Cancer Quality of Life Questionnaire BR-23 | Baseline, 6 months, 12 months
  Participants to complete the EORTC Quality of Life Questionnaire-BR23. The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-BR23 has demonstrated validity and reliability as a quality of life questionnaires specific for breast cancer. The EORTC QLQ-BR23 is a breast-specific module that comprises of 23 questions to assess body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects, breast symptoms, arm symptoms and upset by hair loss. The scoring approach for the QLQ-BR23 is identical to QLQ-C30. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state). The percent change in scores from baseline is assessed at 6 months and 12 months.

SECONDARY OUTCOMES:
Cardiovascular risk factors (tobacco use) | 3 years
  The cardiovascular risk factor of tobacco use will be identified from review of medical history in electronic medical records, and surveys from participants. The proportion of patients enrolled in the study with this risk factor will be summarized descriptively.
Cardiovascular risk factors (family history) | 3 years
  The cardiovascular risk factor of family history will be identified from review of medical history in electronic medical records, and surveys from participants. The proportion of patients enrolled in the study with this risk factor will be summarized descriptively.
Cardiovascular risk factors (hypertension) | 3 years
  The cardiovascular risk factor of hypertension will be identified from review of medical history in electronic medical records, and surveys from participants. The proportion of patients enrolled in the study with this risk factors will be summarized descriptively.
Referrals for individuals with pre-diabetes | 3 years
  Total number of individuals with (prediabetes) referred to established institutional programs and resources. The number of referrals overall, by disease type, and per patient will be summarized descriptively.
Referrals for individuals with diabetes | 3 years
  Total number of individuals with diabetes referred to established institutional programs and resources. The number of referrals overall, by disease type, and per patient will be summarized descriptively.
Referrals for individuals with risk of cardiovascular disease | 3 years
  Total number of individuals with risk factors for cardiovascular disease referred to established institutional programs and resources. The number of referrals by disease type, and per patient will be summarized descriptively.
Prevalence of prediabetes in women with breast cancer versus healthy individuals | 3 years
  Compare the prevalence of prediabetes in women with breast cancer versus healthy controls from a national database, controlling for age and other confounding factors. The investigators will obtain access to a national database that provides information on the incidence of prediabetes, diabetes, hyperlipidemia, and history of breast cancer. The investigators will compare the expected number of incident cases of prediabetes to the observed number in The investigators' cohort, adjusting for age and race.
Prevalence of diabetes in women with breast cancer versus healthy individuals | 3 years
  Prevalence of of diabetes in women with breast cancer versus healthy controls from a national database, controlling for age and other confounding factors. The investigators will obtain access to a national database that provides information on the incidence of prediabetes, diabetes, hyperlipidemia, and history of breast cancer. The investigators will compare the expected number of incident cases of diabetes to the observed number in The investigators' cohort, adjusting for age and race.
Prevalence of hyperlipidemia in women with breast cancer versus healthy individuals | 3 years
  Prevalence of hyperlipidemia in women with breast cancer versus healthy controls from a national database, controlling for age and other confounding factors. The investigators will obtain access to a national database that provides information on the incidence of prediabetes, diabetes, hyperlipidemia, and history of breast cancer. The investigators will compare the expected number of incident cases of hyperlipidemia to the observed number in The investigators cohort, adjusting for age and race.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sheng, M.D., Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No